CLINICAL TRIAL: NCT04273334
Title: Application of 68Ga NEB PET Imaging in the Diagnosis and Evaluation of Lymphatic Disorders, Including Lymphedema, Lymphangioma, Lymphangioleiomyomatosis, Plastic Bronchitis, Lymphadenopathy Caused by Rheumatoid Arthritis, Etc.
Brief Title: Application of 68Ga NEB PET Imaging in the Diagnosis and Evaluation of Lymphatic Disorders
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCH-NM26
Record Dates: First submitted 2020-02-15; First posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Lymphatic Disorders
MeSH Terms: conditions — Lymphatic Diseases | interventions — 68Ga-1,4,7-triazacyclononane-N,N',N''-triacetic acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-NEB injection and PET/CT scan (Experimental): Patients for lymphatic disorders imaging: The patients were subcutaneously injected with 68Ga-NEB and underwent PET/CT scan 20~40min after the injection.
  Interventions: Drug: 68Ga-NEB

INTERVENTIONS:
Drug: 68Ga-NEB — 68Ga-NEB were injected into the patients before the PET/CT scans
  Other Names: 68Ga-NOTA-Even's Blue

SUMMARY:
This is an open-label whole-body PET/CT study for investigating the value of 68Ga NEB PET imaging in the diagnosis and evaluation of lymphatic disorders including lymphedema, lymphangioma, lymphangioleiomyomatosis, plastic bronchitis, lymphadenopathy caused by rheumatoid arthritis, etc.

DETAILED DESCRIPTION:
No fasting, hydration or other specific preparation was requested on the day of imaging.

Patients for lymphatic drainage disorders imaging underwent whole-body PET/CT acquisitions 20-40 min after subcutaneously injected into first and second interdigital spaces of both feet or hands of 74-111 MBq (2-3 mCi) 68Ga-NEB with each bed position lasted for 2 min.

A MIM workstation was used for post-processing. The visual method was used to evaluate the lymphatic system, including the morphology and the distribution of the lymphatic system. Semiquantitative methods were applied for image analysis.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to provide a written informed consent; Males and females, ≥18 years old； Diagnostic CT or MRI suggesting a diagnosis of lymphatic system lesion(s). In suspicion of lymphedema, lymphangioma, lymphangioleiomyomatosis, plastic bronchitis, lymphadenopathy caused by rheumatoid arthritis, etc.

Exclusion Criteria:

* Females planning to bear a child recently or with childbearing potential; Known severe allergy or hypersensitivity to IV radiographic contrast； Inability to lie still for the entire imaging time because of cough, pain, etc. Inability to complete the needed examinations due to severe claustrophobia, radiation phobia, etc.

Concurrent severe and/or uncontrolled and/or unstable other medical disease that, in the opinion of the investigator, may significantly interfere with study compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value of 68Ga NEB in lymphatic lesion | 1 years
  The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake value (SUV) of the tracer in lymphatic lesion will be measured.

SECONDARY OUTCOMES:
Adverse events collection | 1 week
  Adverse events within 1 week after the injection and scanning of patients and patients will be followed and assessed

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD,PhD, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Science and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No